CLINICAL TRIAL: NCT03779633
Title: Preoperative Locally Applied Oestrogen in Postmenopausal Women With Pelvic Organ Prolapse: Changes in Subjective and Objective Outcome - a Prospective, Randomized, Double-blind, Placebo-controlled, Multicenter Study
Brief Title: Preoperative Oestrogen in Postmenopausal Women With Pelvic Organ Prolapse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Barbara Bodner-Adler, Clinical Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EstrogenPOP
Record Dates: First submitted 2018-07-29; First posted 2018-12-19 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: Local Oestrogen
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Double-blind, Placebo-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Linoladiol Estradiol (Experimental): Linoladiol Estradiol cream 6 weeks before surgery of pelvic organ prolapse
  Interventions: Drug: Linoladiol Estradiol
- Placebo (Placebo Comparator): Placebo cream 6 weeks before surgery of pelvic organ prolapse
  Interventions: Other: Placebo vaginal cream

INTERVENTIONS:
Drug: Linoladiol Estradiol — Linoladiol Estradiol Initial dose (week 1): 1 application (2g Linoladiol = 0.2mg Estradiol) every day for the first week Maintenance dose 1 (week 2) : 1 application (2g Linoladiol = 0.2mg Estradiol) every 48 hours the following week.
  Maintenance dose 2 (week 3-6): 1 application (2g Linoladiol = 0.2mg Estradiol) twice per week the following 4 weeks.
  Route of administration: intravaginally by means of a calibrated applicator before retiring at night Duration: 6 weeks
  Other Names: Montavit ATC Code G03CA03
  Arms: Linoladiol Estradiol
Other: Placebo vaginal cream — Initial dose (week 1): 1 application every day for the first week Maintenance dose 1 (week 2) : 1 application every 48 hours the following week.
  Maintenance dose 2 (week 3-6): 1 application twice per week the following 4 weeks.
  Route of administration: intravaginally by means of a calibrated applicator before retiring at night Duration: 6 weeks
  Arms: Placebo

SUMMARY:
Introduction With increasing age the incidence of pelvic organ prolapse (POP) rises and will increase substantially in the future according to forecasting studies. It is possible that oestrogens, alone or in combination with other forms of therapy, may assist in the management of POP by increasing collagen synthesis and thereby improving the strength of the weakened vaginal epithelium. Yet, studies investigating the effect of topical oestrogen and its impact on POP associated symptoms, both self-reported improvement and observations of objective improvement, are lacking.

Objective To evaluate the subjective efficacy concerning prolapse associated complaints measured by the German pelvic floor questionnaire (domain POP: POP-score) after preoperative use of local oestrogen compared to preoperative placebo treatment in postmenopausal women with symptomatic pelvic organ prolapse. Further variables of interest are POP-score after 3 months, differences regarding the objective prolapse quantification system (POP-Q), surgical outcome and tissue operability assessed by the surgeon.

Methods In this prospective, randomized, double-blind, placebo-controlled, multicenter study the investigators aim to include 120 postmenopausal women with symptomatic pelvic organ prolapse and indicated operative procedure. An analysis of covariance will be computed with the depending variable POP-score after 6 weeks and the independent variables group (verum versus placebo) and Pop-Score at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Able to read, understand and sign informed consent
* Able to apply a vaginal cream
* Symptomatic pelvic organ prolapse with planned and indicated prolapse surgical repair

Exclusion Criteria:

* Suspicion or history of breast cancer or other oestrogen responsive malignancies (endometrial cancer)
* unexplained abnormal vaginal bleeding
* history of deep vein thrombosis
* inherited or acquired blood clotting disorders (eg, APC resistance, Antithrombin III deficiency)
* transient ischaemic attack, myo- cardial infarction or ischaemic heart disease
* Hypersensitivity to oestrogen
* Unable to read and sign informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
subjective prolapse associated symptoms (measured with the validated German pelvic floor questionnaire) | change from baseline POP Score at 6 weeks after treatment
  treatment efficacy of preoperative vaginally administered oestrogen in postmenopausal women with symptomatic pelvic organ prolapse in comparison to placebo, measured by a subjective questionnaire. 42 questions. Range 0 to 3 points for each question. Lower values represent a better outcome

SECONDARY OUTCOMES:
operative time in minutes | up to 1 week postoperative
  effect of preoperative vaginally administered oestrogen on postoperative outcome in comparison to placebo
length of stay in days | up to 1 week postoperative
  effect of preoperative vaginally administered oestrogen on postoperative outcome in comparison to placebo
intraoperative blood loss in ml | up to 1 week postoperative
  effect of preoperative vaginally administered oestrogen on postoperative outcome in comparison to placebo
blood circulation of the tissue (good, regular, scarce, no blood circulation) | on day of surgery
  differences in tissue operability between the two groups assessed by means of a questionnaire which is filled in by the surgeon after the operation
separability of the tissue layers (good, regular, scarce, not possible) | on day of surgery
  differences in tissue operability between the two groups assessed by means of a questionnaire which is filled in by the surgeon after the operation
easy separation from the bladder (yes/no) | on day of surgery
  differences in tissue operability between the two groups assessed by means of a questionnaire which is filled in by the surgeon after the operation
easy opening of the Douglas cavity (Yes/no) | on day of surgery
  differences in tissue operability between the two groups assessed by means of a questionnaire which is filled in by the surgeon after the operation
subjective (all domains of the pelvic floor questionnaire) outcome 3 months postoperative | 3 months postoperative
  possible differences regarding subjective outcome parameters between intervention and placebo-group 3 months after operation. 42 questions. Range 0 to 3 points for each question. Lower values represent a better outcome.
objective (POP-Q score) outcome 3 months postoperative | 3 months postoperative
  possible differences regarding objective outcome parameters between intervention and placebo-group 3 months after operation. POP-Q Score (Score between 0 and 4). The POP- quantification system consists of six defined points of measurement (Aa, Ba, C,D,Ap,Bp) and three other landmarks (GH,TVL, PB). Each is measured in centimeters above the hymen (negative number) or below the hymen (positive number).

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Department of Obstetrics and Gynecology, University of Tulln, Tulln
  - Department of General Gynecology and Gynecologic Oncology of the Medical University Vienna, Vienna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weber MA, Kleijn MH, Langendam M, Limpens J, Heineman MJ, Roovers JP. Local Oestrogen for Pelvic Floor Disorders: A Systematic Review. PLoS One. 2015 Sep 18;10(9):e0136265. doi: 10.1371/journal.pone.0136265. eCollection 2015. PMID 26383760
- [Background] Rahn DD, Good MM, Roshanravan SM, Shi H, Schaffer JI, Singh RJ, Word RA. Effects of preoperative local estrogen in postmenopausal women with prolapse: a randomized trial. J Clin Endocrinol Metab. 2014 Oct;99(10):3728-36. doi: 10.1210/jc.2014-1216. Epub 2014 Jun 20. PMID 24947034
- [Derived] Taithongchai A, Johnson EE, Ismail SI, Barron-Millar E, Kernohan A, Thakar R. Oestrogen therapy for treating pelvic organ prolapse in postmenopausal women. Cochrane Database Syst Rev. 2023 Jul 11;7(7):CD014592. doi: 10.1002/14651858.CD014592.pub2. PMID 37431855
- [Derived] European Urogynaecological Association 2021 Annual Meeting | Hybrid Edition. Female Pelvic Med Reconstr Surg. 2022 Apr 1;28(4):244-271. doi: 10.1097/SPV.0000000000001172. No abstract available. PMID 35443258